CLINICAL TRIAL: NCT02643290
Title: Efficacy of Peak Scoliosis Brace in Pain Management For Adult Scoliosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aspen Medical Products (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156_2015bis
Record Dates: First submitted 2015-12-24; First posted 2015-12-31 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Back Pain
Keywords: Adult Scoliosis; Pain Management; Orthosis
MeSH Terms: conditions — Back Pain; Scoliosis; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients (Other): Adult patients with low back pain secondary to an high degree scolisis are treated by fiting with a brace 2-4 hours a day and tracked for 6 months.
  Interventions: Device: Peak Scoliosis Bracing System

INTERVENTIONS:
Device: Peak Scoliosis Bracing System — Brace is fit to adult scoliosis patients for 2-4 hours a day and tracked for six months.

SUMMARY:
Aim of the study is to evaluate a new brace that has become available, the Peak Scoliosis Brace (Aspen Medical Products) designed to alleviate pain for adult patients with chronic pain secondary to scoliosis.

20 adults with back pain secondary to Idiopathic Scoliosis will be recruited. The sample size was calculated considering the data collected during the development of the brace in the US. Patients will be evaluated at baseline immediately before starting with the brace and after 4 weeks and 6 months. The brace must be worn for at least 2-4 hours per day.

At each evaluation they will be asked to fill the questionnaires, to be used as outcome measure of the results.

DETAILED DESCRIPTION:
Background: Some adult scoliosis patients suffer significant back pain and risk increased curvature leading to postural collapse. The main approach for these patients according to the current literature is the surgical one, however, surgery is not without complications, is not appropriate for all patients and certain patients do not choose to undergo surgery. Despite the fact that scoliosis has been estimated to affect up to 68% of the population over 60, there is scant literature about conservative treatments for adult scoliosis; a case report and a case series demonstrated the effectiveness of scoliosis specific exercise to stop progression, while another study reported the effectiveness of a soft brace in reducing pain at short time. Custom fabricated rigid torso braces, similar to those commonly used for children are sometimes used in adult patients, however, the goal of these braces is to correct and/or sustain the sagittal plane of patients, no data have been published on the efficacy of these braces in relief of pain, and such braces are typically not well tolerated by adults. Recently a new brace has become available, the Peak Scoliosis Brace (Aspen Medical Products) designed to alleviate pain for adult patients with chronic pain secondary to scoliosis.

Aim: to test the efficacy of the Peak Scoliosis Brace in reducing pain in adult scoliosis patients.

Study design: prospective cohort study. Population: 20 adults with back pain secondary to Idiopathic Scoliosis. The sample size was calculated considering the data collected during the development of the brace in the US, and the first 2 patients fitted in Italy. Setting alpha at 0.05 and the power at 0.8, with a mean expected improvement of 2 point in the pain NRS, 16 patients would be necessary.

Considering the possibility of 25% drop out the investigators decided to recruit 20 subjects.

Statistical analysis: If data will be normally distributed, the investigators will use a paired t-test. Otherwise, non-parametric statistical tests will be applied.

Protocol: patients will be evaluated at baseline immediately before starting with the brace and after 4 weeks and 6 months. The brace must be worn for at least 2-4 hours per day. At each evaluation they will be asked to fill the NRS, Rolland Morris Questionnaire and COMI.

ELIGIBILITY:
Inclusion Criteria:

* Must have significant back pain from idiopathic or degenerative scoliosis
* Idiopathic or degenerative scoliosis with Cobb angle > 30"
* Age > 18 years

Exclusion Criteria:

* Prior back surgery
* Secondary scoliosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Pain Relief | At start, 4 weeks, 6 months
  Change in pain from baseline will be measured by means of the Core Outcome Measures Index

SECONDARY OUTCOMES:
Pain Relief | At start, 4 weeks, 6 months
  Oswestry Disability Index
Pain Relief | At start, 4 weeks, 6 months
  Roland Morris Disability Questionnaire
Pain Relief | At start, 4 weeks, 6 months
  Numerical Rating Scale

REFERENCES:
- [Derived] Zaina F, Poggio M, Di Felice F, Donzelli S, Negrini S. Bracing adults with chronic low back pain secondary to severe scoliosis: six months results of a prospective pilot study. Eur Spine J. 2021 Oct;30(10):2962-2966. doi: 10.1007/s00586-021-06808-1. Epub 2021 Mar 17. PMID 33733328